CLINICAL TRIAL: NCT04755231
Title: Post-Market Clinical Study of the AcrySof® IQ PanOptix® Presbyopia Correcting Intraocular Lens in a Chinese Population
Brief Title: Post-Market Clinical Study of the PanOptix Intraocular Lens (IOL) in a Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILH297-C004
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Aphakia; Presbyopia
Keywords: Cataract; Intraocular Lens
MeSH Terms: conditions — Aphakia; Presbyopia; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PanOptix IOL (Experimental): AcrySof IQ PanOptix Presbyopia Correcting IOL implanted in the capsular bag in the posterior chamber of the eye during cataract surgery
  Interventions: Device: AcrySof IQ PanOptix Presbyopia Correcting IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: AcrySof IQ PanOptix Presbyopia Correcting IOL — UV and blue-light filtering foldable multifocal IOL with a +2.17 diopter (D) addition power of intermediate visual acuity and a +3.25 D addition power of near visual acuity. This device is approved in China.
  Other Names: Model TFNT00
Procedure: Cataract surgery — Cataract extraction by phacoemulsification, followed by implantation of the AcrySof IQ PanOptix Presbyopia Correcting IOL

SUMMARY:
The primary objective of this clinical study is to assess the clinical performance of the PanOptix IOL in a Chinese population.

DETAILED DESCRIPTION:
In this clinical study, subjects will be implanted with the PanOptix IOL in both eyes. The second eye surgery will occur 7-28 days after the first eye. A total of 11 scheduled visits are planned, including a screening visit, two operative visits, and 8 postoperative visits. The total expected duration of the subject's participation will be about 14 months. This study will be conducted in China.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to comprehend and sign an informed consent form;
* Able to complete all study visits required in the protocol;
* Chinese; diagnosed with cataracts in both eyes;
* Planned bilateral cataract removal by routine phacoemulsification;
* Pre-operative regular corneal astigmatism of less than 1.0 diopter (D);
* Pre-operative best corrected distance visual acuity (BCDVA) worse than or equal to 0.3 LogMAR in each eye;
* Potential postoperative best corrected distance visual acuity (BCDVA) of 0.3 logMAR or better in both eyes based on the investigator expert medical opinion.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Glaucoma, diabetic retinopathy, retinitis pigmentosa and any pathologic changes associated with the optic nerve;
* Clinically significant corneal diseases;
* Clinically significant/severe dry eye that would affect study measurements based on the investigator's expert medical opinion;
* Previous intraocular or corneal surgery;
* Pregnancy or lactation during study or planning to be pregnant/lactating;
* Systemic medications that, in the opinion of the Investigator, may confound the outcome or increase the risk to the subject;
* Other planned ocular surgical procedures;
* Patients who desire monovision correction.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Project Manager, Surgical, Study Director — Alcon (China) Ophthalmic Product Co., Ltd.
Locations (9):
- China (9):
  - Peking University People's Hospital, Beijing
  - Beijing Tongren Hospital Capital Medical University, Beijing
  - Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guandong
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Ophthalmic Hospital Affiliated to Shandong University of Traditional Chinese Medicine, Shandong
  - Eye & ENT Hospital of Fudan University, Shanghai
  - Shanxi Eye Hospital, Shanxi
  - West China Hospital of Sichuan University, Sichuan
  - Tianjin Medical University Eye Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 9 investigative sites located in China.
Pre-assignment Details: Of the 181 who signed an informed consent document, 37 participants were discontinued prior to implantation: 27 participants were screen failures, and 10 participants withdrew. This reporting group includes all participants with attempted implantation (144).
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | PanOptix IOL
Started | 144; 288 eyes
Attempted Implantation, First Eye | 144; 144 eyes
Attempted Implantation Second Eye | 142; 142 eyes
Successful Implantation, First Eye | 144; 144 eyes
Successful Implantation Second Eye | 142; 142 eyes
Completed | 134; 268 eyes
Not Completed | 10; 20 eyes
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: This analysis population includes all subjects who had successful IOL implantation in at least one eye and at least one postoperative effectiveness assessment.
Arm/Group | PanOptix IOL
Number analyzed (Participants) | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (9.19)
Age, Customized [Count of Participants; unit: Participants]
  Less than 65 years | 72
  65 years and older | 72
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese/Asian | 144
Region of Enrollment [Count of Participants; unit: Participants]
  China | 144

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Best Corrected Distance Visual Acuity (BCDVA) Equal to or Better Than 0.3 LogMAR - Monocular
Description: Visual acuity (VA) was assessed monocularly (eyes individually) with best refractive correction in place under photopic (well-lit) conditions at a distance of 5 meters using Chinese Standard Logarithmic VA charts. LogMAR typically ranges from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision). Lower scores indicate better vision. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Month 6 (180-210 days post second eye surgery, 187-238 days post first eye surgery)
Population: Full Analysis Set with data at visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- PanOptix IOL - First Eye; PanOptix IOL - Second Eye; PanOptix IOL - All Eyes: AcrySof IQ PanOptix Presbyopia Correcting IOL implanted in the capsular bag in the posterior chamber of the eye during cataract surgery
Arm/Group | PanOptix IOL - First Eye | PanOptix IOL - Second Eye | PanOptix IOL - All Eyes
Number analyzed (Participants) | 135 | 135 | 135
Number analyzed (eyes) | 135 | 135 | 270
percentage of eyes | 100 | 98.5 | 99.3

2. Primary Outcome: Percentage of Eyes With Best Corrected Distance Visual Acuity (BCDVA) Equal to or Better Than 0.3 LogMAR - Binocular
Description: VA was assessed binocularly (eyes together) with best refractive correction in place under photopic conditions at a distance of 5 meters using Chinese Standard Logarithmic VA charts. LogMAR typically ranges from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision). Lower scores indicate better vision. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Month 6 (180-210 days post second eye surgery, 187-238 days post first eye surgery)
Population: Full Analysis Set with data at visit
Measure: Number; unit: percentage of participants
Units Other Than Participants: eyes
Arm/Group | PanOptix IOL
Number analyzed (Participants) | 135
Number analyzed (eyes) | 270
percentage of participants | 100

3. Primary Outcome: Mean Best Corrected Distance Visual Acuity (BCDVA) - Monocular
Description: as for outcome 1
Time Frame: Month 6 (180-210 days post second eye surgery, 187-238 days post first eye surgery)
Population: Full Analysis Set with data at visit
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | PanOptix IOL - First Eye | PanOptix IOL - Second Eye | PanOptix IOL - All Eyes
Number analyzed (Participants) | 135 | 135 | 135
Number analyzed (eyes) | 135 | 135 | 270
logMAR | -0.02 (0.102) | -0.02 (0.119) | -0.02 (0.110)

4. Primary Outcome: Mean Best Corrected Distance Visual Acuity (BCDVA) - Binocular
Description: as for outcome 2
Time Frame: Month 6 (180-210 days post second eye surgery, 187-238 days post first eye surgery)
Population: Full Analysis Set with data at visit
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | PanOptix IOL
Number analyzed (Participants) | 135
Number analyzed (eyes) | 270
logMAR | -0.08 (0.102)

5. Primary Outcome: Mean Distance Corrected Intermediate Visual Acuity (DCIVA) - Monocular
Description: VA was assessed monocularly (eyes individually) with distance correction in place (plus or minus power) under photopic conditions at a distance of 60 centimeters using Chinese Standard Logarithmic VA charts. LogMAR typically ranges from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision). Lower scores indicate better vision. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Month 6 (180-210 days post second eye surgery, 187-238 days post first eye surgery)
Population: Full Analysis Set with data at visit
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | PanOptix IOL - First Eye | PanOptix IOL - Second Eye | PanOptix IOL - All Eyes
Number analyzed (Participants) | 135 | 135 | 135
Number analyzed (eyes) | 135 | 135 | 270
logMAR | 0.073 (0.1110) | 0.072 (0.1329) | 0.073 (0.1222)

6. Primary Outcome: Mean Distance Corrected Intermediate Visual Acuity (DCIVA) - Binocular
Description: VA was assessed binocularly (eyes together) with distance correction in place (plus or minus power) under photopic conditions at a distance of 60 centimeters using Chinese Standard Logarithmic VA charts. LogMAR typically ranges from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision). Lower scores indicate better vision. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Month 6 (180-210 days post second eye surgery, 187-238 days post first eye surgery)
Population: Full Analysis Set with data at visit
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | PanOptix IOL
Number analyzed (Participants) | 135
Number analyzed (eyes) | 270
logMAR | 0.018 (0.0875)

7. Primary Outcome: Mean Distance Corrected Near Visual Acuity (DCNVA) - Monocular
Description: VA was assessed monocularly (eyes individually) with distance correction in place (plus or minus power) under photopic conditions at a distance of 40 centimeters using Chinese Standard Logarithmic VA charts. LogMAR typically ranges from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision). Lower scores indicate better vision. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Month 6 (180-210 days post second eye surgery, 187-238 days post first eye surgery)
Population: Full Analysis Set with data at visit
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | PanOptix IOL - First Eye | PanOptix IOL - Second Eye | PanOptix IOL - All Eyes
Number analyzed (Participants) | 135 | 135 | 135
Number analyzed (eyes) | 135 | 135 | 270
logMAR | 0.082 (0.1074) | 0.078 (0.1175) | 0.080 (0.1124)

8. Primary Outcome: Mean Distance Corrected Near Visual Acuity (DCNVA) - Binocular
Description: VA was assessed binocularly (eyes together) with distance correction in place (plus or minus power) under photopic conditions at a distance of 40 centimeters using Chinese Standard Logarithmic VA charts. LogMAR typically ranges from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision). Lower scores indicate better vision. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Month 6 (180-210 days post second eye surgery, 187-238 days post first eye surgery)
Population: Full Analysis Set with data at visit
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | PanOptix IOL
Number analyzed (Participants) | 135
Number analyzed (eyes) | 270
logMAR | 0.025 (0.0865)

9. Primary Outcome: Number of Ocular Treatment Emergent Adverse Events
Description: An adverse event was defined as any adverse medical event that occurred during the clinical trial whether or not it was related to the investigational medical device or test procedure. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Month 12 (360-390 days post second eye surgery, 367-418 days post first eye surgery)
Population: Safety Analysis Set: All subjects/eyes with attempted implantation with the test article (successful or aborted after contact with the eye).
Measure: Number; unit: adverse events
Units Other Than Participants: eyes
Arm/Group | PanOptix IOL - First Eye | PanOptix IOL - Second Eye | PanOptix IOL - All Eyes
Number analyzed (Participants) | 144 | 142 | 144
Number analyzed (eyes) | 144 | 142 | 286
adverse events | 37 | 33 | 70

10. Primary Outcome: Number of Non-Ocular Treatment Emergent Adverse Events
Description: as for outcome 9
Time Frame: Month 12 (360-390 days post second eye surgery, 367-418 days post first eye surgery)
Population: as for outcome 9
Measure: Number; unit: adverse events
Groups:
- Pan Optix IOL: AcrySof IQ PanOptix Presbyopia Correcting IOL implanted in the capsular bag in the posterior chamber of the eye during cataract surgery
Arm/Group | Pan Optix IOL
Number analyzed (Participants) | 144
adverse events | 28

11. Primary Outcome: Number of Secondary Surgical Interventions
Description: A secondary surgical intervention (SSI) was defined as a surgical procedure occurring after primary implantation of the IOL. Posterior capsulotomies were excluded from the definition of secondary surgical interventions. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Month 12 (360-390 days post second eye surgery, 367-418 days post first eye surgery)
Population: as for outcome 9
Measure: Number; unit: secondary surgical interventions
Units Other Than Participants: eyes
Arm/Group | PanOptix IOL - First Eye | PanOptix IOL - Second Eye | PanOptix IOL - All Eyes
Number analyzed (Participants) | 144 | 142 | 144
Number analyzed (eyes) | 144 | 142 | 286
secondary surgical interventions | 0 | 0 | 0

12. Primary Outcome: Number of Participants Reporting a Severe Visual Disturbance (QUVID)
Description: The Questionnaire for Visual Disturbances (QUVID) is a patient-reported outcomes questionnaire that collects responses about 7 vision-related experiences. For each experience, the participant was asked, "In the Past 7 Days, How Severe Was Your Worst Experience" and responded on a 5-point scale, where 0-4 scale, where 0=none, 1=a little, 2=mild, 3=moderate, and 4=severe. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Month 6 (180-210 days post second eye surgery, 187-238 days post first eye surgery); Month 12 (360-390 days post second eye surgery, 367-418 days post first eye surgery)
Population: Safety Analysis Set with data at visit
Measure: Number; unit: participants
Groups:
- Month 6 Post Second Eye Implantation; Month 12 Post Second Eye Implantation: AcrySof IQ PanOptix Presbyopia Correcting IOL implanted in the capsular bag in the posterior chamber of the eye during cataract surgery
Arm/Group | Month 6 Post Second Eye Implantation | Month 12 Post Second Eye Implantation
Number analyzed (Participants) | 135 | 135
participants
  Starbursts | 13 | 21
  Halos | 9 | 6
  Glare: number analyzed (Participants) | 135 | 133
  Glare | 6 | 3
  Hazy Vision | 3 | 1
  Blurred Vision | 3 | 2
  Double Vision: number analyzed (Participants) | 133 | 129
  Double Vision | 0 | 0
  Dark Area: number analyzed (Participants) | 135 | 134
  Dark Area | 0 | 0

13. Primary Outcome: Number of Participants Reporting a Most Bothersome Visual Disturbance (QUVID)
Description: The Questionnaire for Visual Disturbances (QUVID) is a patient-reported outcomes questionnaire that collects responses about 7 vision-related experiences. For each experience, the participant was asked, "In the Past 7 Days, How Much Were You Bothered With" and responded on a 5-point scale, where 0=not bothered at all, 1=bothered a little, 2=bothered somewhat, 3=bothered quite a bit, and 4=bothered very much (most bothersome). No hypothesis testing was pre-specified for this endpoint.
Time Frame: as for outcome 12
Population: Safety Analysis Set with data at visit
Measure: Number; unit: participants
Arm/Group | Month 6 Post Second Eye Implantation | Month 12 Post Second Eye Implantation
Number analyzed (Participants) | 135 | 135
participants
  Starbursts | 2 | 2
  Halos | 3 | 2
  Glare: number analyzed (Participants) | 135 | 133
  Glare | 4 | 2
  Hazy Vision | 0 | 0
  Blurred Vision | 1 | 1
  Double Vision: number analyzed (Participants) | 135 | 129
  Double Vision | 0 | 0
  Dark Area: number analyzed (Participants) | 135 | 134
  Dark Area | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of enrollment until study exit, approximately 14 months.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for Pretreatment and Systemic AEs is reported in units of subjects. "At Risk" population for Ocular AEs is reported in units of eyes. This analysis population includes all subjects/eyes with attempted implantation with the test article (successful or aborted after contact with the eye).
Groups:
- Pretreatment: Events reported in this group occurred prior to attempted implantation with the test article and may include ocular events in the second eye prior to implantation, as well as overall systemic events.
- PanOptix IOL Ocular - First Eye: Events reported in this group occurred after attempted implantation with the test article and include ocular events in the first implanted eye
- PanOptix IOL Ocular - Second Eye: Events reported in this group occurred after attempted implantation with the test article and include ocular events in the second implanted eye
- PanOptix IOL Systemic: Events reported in this group occurred after attempted implantation with the test article
Arm/Group | Pretreatment | PanOptix IOL Ocular - First Eye | PanOptix IOL Ocular - Second Eye | PanOptix IOL Systemic
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/144 | 0/142 | 0/144
Serious Adverse Events (participants affected / at risk) | 0/144 | 2/144 | 3/142 | 6/144
Other Adverse Events (participants affected / at risk) | 2/144 | 15/144 | 11/142 | 0/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=144) | PanOptix IOL Ocular - First Eye (N=144) | PanOptix IOL Ocular - Second Eye (N=142) | PanOptix IOL Systemic (N=144)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Cystoid macular oedema (Eye disorders) | 0 | 2 | 3 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=144) | PanOptix IOL Ocular - First Eye (N=144) | PanOptix IOL Ocular - Second Eye (N=142) | PanOptix IOL Systemic (N=144)
Dry eye (Eye disorders) | 2 | 15 | 11 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT04755231/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT04755231/SAP_001.pdf